CLINICAL TRIAL: NCT01302873
Title: A Multicenter, Randomized, Double-blind, Placebo- Controlled, Cross-over, Proof of Concept Study Comparing the Effects of Both Single Dose and Repeated Dosing Treatment for 2 Weeks of BGG492 in Patients With Chronic Subjective Tinnitus
Brief Title: Study of BGG492 in Patients With Chronic Subjective Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBGG492A2210; 2010-022166-27 (EudraCT Number)
Record Dates: First submitted 2011-02-07; First posted 2011-02-24 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Chronic Subjective Tinnitus
Keywords: Tinnitus; AMPA Receptor antagonist
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- BGG492 (Experimental)
  Interventions: Drug: BGG492A
- Placebo (Placebo Comparator)
  Interventions: Drug: BGG492A

INTERVENTIONS:
Drug: BGG492A
  Arms: BGG492
Drug: BGG492A
  Arms: Placebo

SUMMARY:
This study will assess the efficacy of a two week treatment with BGG492 in patients with chronic subjective Tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with THI (Tinnitus Handicap Inventory) severity grade 3, 4 or 5 (moderate, severe or catastrophic), chronic (> 6 months and < 36 months) subjective tinnitus
* Willing to abstain from activities that require focused attention, e.g. driving a car or other vehicles, operating machines or engaging in potentially dangerous activities that require focused attention and intact physical balance
* Willing and able to refrain from engaging in activities or work involving loud noise exposure

Exclusion Criteria:

* Patients diagnosed with tinnitus of THI severity grade equal to 2 or 1
* Patients with diagnosis of intermittent or pulsatile tinnitus
* Patients who have tinnitus as a concomitant symptom of a treatable otological disease (such as otitis media, Menière's disease, otosclerosis), neurological tumors or/and have temporo-mandibular joint disorders
* Patients with a history of frequent middle ear infections (> 3 infections per year during the last 3 years)
* Patients with diagnosed anxiety disorders, depression, schizophrenia or other significant psychiatric diseases requiring current drug treatment or patients who required treatment in the previous 3 months for these diseases.
* Patients with current unilateral or bilateral hearing loss of 75 dB or more in one or more tested frequencies (125 Hz, 250 Hz, 1 kHz, 2 kHz, 4 kHz, 6 kHz, 8 kHz)
* Patients with Vestibular Schwannoma
* Patients with a cochlear implant
* Patients with regular intake of central nervous system acting drugs for the treatment of tinnitus in the previous 6 months prior to initial dosing

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in tinnitus loudness using a visual analogue scale (VAS) | after 15 days of treatment
Change in Clinical status of tinnitus (patients' reaction to tinnitus) using the TBF-12 (Tinnitus Impairment Questionnaire) | after 15 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Lepzig
- Novartis Investigative Site, Groningen, Netherlands

REFERENCES:
- [Derived] Kucher K, Johns D, Wagner F, Abd-Elaziz K, Derne C, Sverdlov O, Pfister CU, Langguth B. Efficacy and safety of single- and repeated-selurampanel dosing for 2 weeks in patients with chronic subjective tinnitus: Results of a randomized, double-blind, placebo-controlled, cross-over, proof-of-concept phase IIa study. Prog Brain Res. 2021;260:423-440. doi: 10.1016/bs.pbr.2020.12.004. Epub 2021 Jan 20. PMID 33637230